CLINICAL TRIAL: NCT04105504
Title: Oral Glutathione As A Skin Whitening Agent: A Randomized, Double-Blind, Placebo-Controlled Multicenter Clinical Trial
Brief Title: Oral Glutathione As A Skin Whitening Agent
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr Irma Bernadette S Sitohang (Other)
Responsible Party: Sponsor-Investigator, Dr Irma Bernadette S Sitohang, Dr. dr. Irma Bernadette S. Sitohang, SpKK(K) - Head of Cosmetic Dermatology Division of Dermatology and Venereology Department of Faculty of Medicine Universitas Indonesia / Cipto Mangunkusumo Hospital, Rumah Sakit Pusat Angkatan Darat Gatot Soebroto
Organization: Rumah Sakit Pusat Angkatan Darat Gatot Soebroto (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCTGlutathione
Record Dates: First submitted 2019-08-08; First posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Glutathione; Skin Whitening
Keywords: glutathione; whitening
MeSH Terms: interventions — Glutathione

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glutathione Group (Experimental): Subjects were randomised to receive Glutathione capsules. The capsules were taken once daily for 12 weeks and evaluated every 4 weeks.
  Interventions: Drug: Glutathione
- Placebo Group (Placebo Comparator): Subjects were randomised to receive Placebo capsules, which were identical in appearance and packaged in identical-looking containers with the Glutathione capsules. The capsules were taken once daily for 12 weeks and evaluated every 4 weeks.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Glutathione — Oral glutathione capsule (500 mg), were taken once daily by the subjects.
  Other Names: L-Gluthatione
  Arms: Glutathione Group
Drug: Placebo oral tablet — Placebo oral capsule were taken once daily by the subjects.
  Arms: Placebo Group

SUMMARY:
The objective of the study was to evaluate the efficacy and safety of oral glutathione for 12 weeks, used as a skin-whitening agent. The study was a randomized, double-blind, placebo-controlled, multicenter study, set at Dermatology outpatient clinic at three different hospitals in Indonesia, Gatot Seobroto Army Hospital Jakarta, Dr. dr. Wahiddin Soedirohoesodo Hospital Makassar, and University of Sumatera Utara Teaching Hospital Medan. Ninety healthy females, aged between 33 and 50 years, were randomized to receive either glutathione capsules or placebo for 12 weeks and evaluated every 4 weeks. The main outcome was total reduction (improvement) of spot UV, spot polarization, and skin tone measured at five different sites for each indices, recorded by Janus Facial Analysis System®.

DETAILED DESCRIPTION:
The objective of the study was to evaluate the efficacy and safety of oral glutathione for 12 weeks, used as a skin-whitening agent.

The study was a randomized, double-blind, placebo-controlled, multicenter study, set at Dermatology outpatient clinic at three different hospitals in Indonesia, Gatot Seobroto Army Hospital Jakarta, Dr. dr. Wahiddin Soedirohoesodo Hospital Makassar, and University of Sumatera Utara Teaching Hospital Medan.

Ninety healthy females, aged between 33 and 50 years, were randomized to receive either glutathione capsules (500 mg) or placebo capsules, which were identical in appearance and packaged in identical-looking containers. The capsules were taken once daily for 12 weeks and evaluated every 4 weeks. Compliance was assessed by counting the remaining capsules at each follow-up visit.

At each follow-up visit, subjects were asked to grade the overall response and questioned regarding adverse events. The objective or main outcome was total reduction (improvement) of spot UV, spot polarization, and skin tone measured at five different sites for each indices, recorded by Janus Facial Analysis System®.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with skin type Fitzpatrick IV and V
* Women aged from 30 to 55 years with an understanding of all the information given by a written consent form
* Working indoor office jobs (for minimum 8 hours)

Exclusion Criteria:

* Personal or family history of skin cancer, especially melanoma
* Consumption of any preparations containing glutathione within 1 month of enrollment
* Use of any topical skin brightening or whitening preparations within 1 month of enrollment
* Pigmentary disorders or any dermatoses, which may affect the measurement within the study areas
* A pregnant or breastfeeding mother
* Personal history of drug allergy or skin disorder due to side effects of oral therapy

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-04-08 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Spot UV at 4 weeks | 4 weeks
  Total reduction (improvement) of spot UV
Change from Baseline Spot Polarization at 4 weeks | 4 weeks
  Total reduction (improvement) of spot polarization
Change from Baseline Skin Tone at 4 weeks | 4 weeks
  Improvement of skin tone
Change from Baseline Spot UV at 8 weeks | 8 weeks
  Total reduction (improvement) of spot UV
Change from Baseline Spot Polarization at 8 weeks | 8 weeks
  Total reduction (improvement) of spot polarization
Change from Baseline Skin Tone at 8 weeks | 8 weeks
  Improvement of skin tone
Change from Baseline Spot UV at 12 weeks | 12 weeks
  Total reduction (improvement) of spot UV
Change from Baseline Spot Polarization at 12 weeks | 12 weeks
  Total reduction (improvement) of spot polarization
Change from Baseline Skin Tone at 12 weeks | 12 weeks
  Improvement of skin tone

SECONDARY OUTCOMES:
Subjective Improvement at 4 weeks | 4 weeks
  Subjects were asked to grade the overall response using rating scale with a multiple-choice question:
  1. minimal improvement
  2. moderate improvement
  3. good improvement
  4. excellent improvement
  Note: The higher improvement represents a better outcome.
Adverse events at 4 weeks | 4 weeks
  Adverse events related to therapy
Subjective Improvement at 8 weeks | 8 weeks
  Subjects were asked to grade the overall response using rating scale with a multiple-choice question:
  1. minimal improvement
  2. moderate improvement
  3. good improvement
  4. excellent improvement
  Note: The higher improvement represents a better outcome.
Adverse events at 8 weeks | 8 weeks
  Adverse events related to therapy
Subjective Improvement at 12 weeks | 12 weeks
  Subjects were asked to grade the overall response using rating scale with a multiple-choice question:
  1. minimal improvement
  2. moderate improvement
  3. good improvement
  4. excellent improvement
  Note: The higher improvement represents a better outcome.
Adverse events at 12 weeks | 12 weeks
  Adverse events related to therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Universitas Indonesia, Jakarta Pusat, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sitohang IBS, Anwar AI, Jusuf NK, Arimuko A, Norawati L, Veronica S. Evaluating Oral Glutathione Plus Ascorbic Acid, Alpha-lipoic Acid, and Zinc Aspartate as a Skin-lightening Agent: An Indonesian Multicenter, Randomized, Controlled Trial. J Clin Aesthet Dermatol. 2021 Jul;14(7):E53-E58. Epub 2021 Jul 1. PMID 34840651